CLINICAL TRIAL: NCT06899646
Title: Safety and Efficacy of BTL-699-2 for Improvement of Mental Well-being
Brief Title: EXOMIND (BTL-699-2) for Improvement of Mental Well-being
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BTL Industries Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BTL-699_CTUS100
Record Dates: First submitted 2025-03-26; First posted 2025-03-28 (Actual); Last update posted 2025-07-21 (Actual); Status verified 2025-03

CONDITIONS: Well-Being, Psychological
Keywords: well-being; TMS; rTMS; ExoTMS; EXOMIND
MeSH Terms: conditions — Psychological Well-Being | interventions — Therapeutics

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Treatment with BTL-699-2 (Experimental): Transcranial magnetic stimulation treatments with the BTL-699-2 device
  Interventions: Device: Treatment with BTL-699-2

INTERVENTIONS:
Device: Treatment with BTL-699-2 — Four transcranial magnetic stimulation treatments with the BTL-699-2 device will be delivered over the left dorsolateral prefrontal cortex, spaced 5 to 10 days apart. The intensity will be adjusted according to the subject's feedback, up to 100% of the individual's motor threshold.
  Other Names: EXOMIND (BTL-699-2) Treatment

SUMMARY:
The goal of this clinical trial is to evaluate if the treatment with EXOMIND (BTL-699-2) device is able to improve mental well-being in adults above the age of 22 years. The main question it aims to answer is:

Does the treatment with EXOMIND (BTL-699-2) device improve mental well-being?

Participants will be asked to:

* Undergo four treatments
* Complete the Warwick Edinburgh Mental Well-being Scale
* Complete the Therapy Comfort Questionnaire
* Complete the Subject Satisfaction & Mental Wellness Questionnaire

DETAILED DESCRIPTION:
The study uses a multi-center, single-arm, open-label, interventional study design. The subjects will be enrolled and assigned to one experimental study arm. All enrolled participants will receive four treatment visits, 5-10 days apart.

The Warwick Edinburgh Mental Well-being Scale (WEMWBS) will be administered to the subjects before the first treatment, after the last treatment, and at the two follow-up visits- 1 month and 3 months after the final session.

The Therapy Comfort Questionnaire will be administered after the last treatment, while the Subject Satisfaction & Mental Wellness Questionnaire will be given after the last treatment and at both follow-up visits.

The total expected duration of subject participation, from the baseline visit to study completion, is approximately five months.

ELIGIBILITY:
Inclusion Criteria:

* Age > 22 years
* Ability to determine the motor threshold of the participant. The participant's motor threshold could be established as the minimum stimulus required to induce contraction of the right thumb
* Subjects willing and able to abstain from partaking in any treatments other than the pre-procedure therapy regime for the improvement of mental well-being, including non-invasive brain stimulation treatments other than the study procedure during study participation
* Willingness to comply with study instructions and to return to the clinic for the required visits
* Women of child-bearing potential* are required to use birth control measures during the whole duration of the study
* If applicable, subjects will be maintained on pre-study psychotherapeutic regime, and neuropsychiatric prescribed medications (including SSRI or other medication) at a stable therapeutic dosage for at least 2 months prior to study entry

Exclusion Criteria:

* Electronic implants (Implanted stimulator devices in or near the head - rTMS devices are contraindicated for use in patients who have active or inactive implants (including device leads), deep brain stimulators, cochlear implants, ocular implant, and vagus nerve stimulators, implanted devices such as cardiac pacemakers, defibrillators, neurostimulators. Contraindicated use could result in serious injury or death.
* Metallic, conductive, ferromagnetic or other magnetic sensitive implants/objects in the head or within 30 cm of the treatment coil (examples include implanted electrodes/stimulators, aneurysm clips or coils, stents, bullet fragments, jewelry and hair barrettes) with some exceptions in the mouth as standard amalgam dental fillings, single post dental implants, and dental bridge work. Failure to follow this restriction could result in serious injury or death.
* Drug pump(s)
* Application in the heart area
* Persons with a tendency to seizure (hypotonic, epileptic), or a personal history of epilepsy
* Ongoing anticoagulation therapy
* Ongoing severe or life-threatening condition
* Pulmonary insufficiency
* Heart disorders
* Renal insufficiency
* Decompensated* hemorrhagic conditions, blood coagulation disorders, cardiovascular diseases
* Malignant or benign tumor
* Fever
* Ongoing pregnancy or nursing
* Ongoing intake disorders such as bulimia or anorexia
* Diagnosis of post-traumatic stress disorder, psychotic disorder or current psychotic symptoms, bipolar disorder, obsessive-compulsive disorder, borderline personality disorder
* Personal history of syncope (except the reflex syncope)
* Vascular, traumatic, tumoral, infectious, or metabolic lesion of the brain, even without a history of seizure, and without anticonvulsant medication
* Withdrawal from one of the following drugs could form a relative hazard for the application of rTMS due to the resulting significant seizure threshold lowering potential: (e.g. alcohol, barbiturates, benzodiazepines, meprobamate, chloralhydrate etc.)
* Systemic infection
* Patients with a broad range of neuropsychiatric diseases are at elevated risk for seizures. Essentially all neurologic conditions with structural cerebral damage (e.g. stroke, multiple sclerosis, traumatic brain injury, Alzheimer's and other neurodegenerative diseases, meningoencephalitis or intracerebral abscess, parenchymal or leptomeningeal cancers)
* History of hyponatremia, hypocalcemia, hypomagnesemia, hypoglycemia, hyperglycemia, renal failure/uremia, liver failure
* History of tendency for raised blood concentrations of pro-convulsant medications due to reduced clearance
* Immunosuppressive therapy with cyclosporine, tacrolimus and other agents that can cause the posterior reversible leukoencephalopathy syndrome
* The use of methamphetamine, barbiturates, cocaine metabolites, opiates and phencyclidine 72 hours before the therapy
* Contradictions for the testing used in the trial, for example, the motor threshold cannot be found or quantified.

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2024-07-08 (Actual); Primary Completion 2025-02-03 (Actual); Study Completion 2025-02-03 (Actual)

PRIMARY OUTCOMES:
Assessment of Change in Mental Well-Being | 15 months
  The change in the score obtained from the Warwick Edinburgh Mental Well-being Scale will be recorded. The questionnaire will be administered at the baseline visit, after the last treatment, at the 1-month and 3-month follow-up visits. The score ranges from 14 to 70 and higher scores indicate greater mental well-being. An improvement is defined as an increase in score.

SECONDARY OUTCOMES:
Assessment of Therapy Comfort | 15 months
  Therapy Comfort questionnaire will be used for evaluating the comfort during the treatment sessions. The Therapy Comfort questionnaire will be administered after the last treatment. Therapy Comfort questionnaire consists of the question "I found the treatment comfortable", to which responses are based on a 5-point Likert scale (1 = "strongly disagree", and 5 = "strongly agree") and the 10-point Numeric Analog Scale for pain (0 = no pain, 10 = worst possible pain"). A higher score for the statement "I found the treatment comfortable", and lower score on the Numeric Analog Scale for pain indicate higher therapy comfort.
Assessment of Satisfaction | 15 months
  Subject Satisfaction with treatment outcomes will be assessed using 5-point Likert Scale Subjects Satisfaction & Mental Wellness questionnaire. The questionnaire will be administered after the last treatment, at the 1-month and 3-month follow-up visits. Responses to questions about satisfaction with the treatment outcomes will range from "strongly disagree" (1 point) to "strongly agree" (5 points). A higher score for each statement indicate better outcomes.
Incidence of Treatment-related Adverse Events | 15 months
  Monitoring of adverse reactions and side effects will be performed for the evaluation of safety of the treatment with the BTL-699-2 device for the improvement of well-being and to identify side effects and adverse events associated with the study treatment.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Contour Medical, Gilbert, Arizona
  - Luxury Psychiatry Medical and Spa, Winter Garden, Florida
  - Yael Halaas, M.D., F.A.C.S., New York, New York